CLINICAL TRIAL: NCT03682796
Title: Phase 1, Multicenter, Open-Label Study of the Antibody-Drug Conjugate TRPH-222 in Subjects With Relapsed and/or Refractory B-Cell Lymphoma
Brief Title: Study of TRPH-222 in Patients With Relapsed and/or Refractory B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Triphase Research and Development III Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TRPH-222-100
Record Dates: First submitted 2018-09-20; First posted 2018-09-25 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Lymphoma; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Lymphoma, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular
Keywords: Antibody-Drug Conjugate; ADC; CD22; SMARTag™ technology; TRPH-222
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escalation (Experimental): Estimated to be <31 subjects across multiple centers
  Interventions: Drug: TRPH-222
- Expansion (Experimental): Estimated to be <121 subjects across multiple centers
  Interventions: Drug: TRPH-222

INTERVENTIONS:
Drug: TRPH-222 — administered by IV, 21-day Cycle

SUMMARY:
This is a Phase 1, multi-center, open-label study of TRPH-222 monotherapy in subjects with relapsed and/or refractory B-cell NHL. The study will be conducted in two Stages: Dose-Escalation, Dose-Expansion.

DETAILED DESCRIPTION:
In Dose Escalation, patients with DLBCL, FL (including transformed FL), MZL, and MCL were to be enrolled per dose cohort. In Dose Expansion, additional response-evaluable patients were to be enrolled in NHL subtype-specific cohorts including DLBCL and FL to confirm the RP2D identified in Escalation. Each stage consisted of screening, baseline, treatment, and follow-up periods. During the treatment period, patients were to be treated indefinitely in 21 day cycles. The EOT assessments were to occur 28 and 60 days after the last study treatment.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years at the time of signing the informed consent
* Histologically confirmed (2016 WHO lymphoma classification) B-cell NHL that is DLBCL, FL (including transformed FL), MZL, or MCL
* Relapsed and/or refractory NHL requiring systemic therapy and have failed, are intolerant to, or are considered ineligible for standard of care anticancer treatments that are known to be potentially curative. Subjects must not be current candidates for HSCT. Participants who refuse standard treatments may also be considered provided that documentation is provided that the subject has been made aware of all therapeutic options
* Eastern Cooperative Oncology Group (ECOG) status 0-2

Exclusion Criteria

* Presence of a leukemic phase of the lymphoma
* "Double hit" or "triple hit" germinal center B cell lymphoma
* Previous solid organ allograft (except for corneal transplant)
* Peripheral neuropathy > NCI-CTCAE Grade 1
* Significant organ dysfunction that would preclude study participation
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias
* Any other serious active disease or co-morbid medical condition, according to the Investigator's decision or Medical Monitor, that will substantially increase the risk associated with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 21 days
  To determine the MTD of TRPH-222

SECONDARY OUTCOMES:
Evaluate incidence and severity of AEs, serious AEs, TRPH-222-related AEs, AEs leading to death or discontinuation from treatment | Up to 28 days after last dose of study drug
  Safety
Tumor Activity | Up to 2 years
  Assess tumor response - ORR for each NHL subtype using Lugano criteria, PFS from first dose to disease progression, OS from first dose to death, DOR for each NHL subtype assessed by Lugano
TRPH-222 Pharmacokinetics (PK) | Each Cycle is 21 days. Days 1, 8, 15 of Cycle 1; Day 1 of Cycle 2 and Cycle 3; Day 1 of every third cycle thereafter; up to Day 28 after last dose of study drug; Day 60 after last dose of study drug
  Maximum concentration of TRPH-222 (Cmax), time to Cmax, Half-life (t 1/2), Exposure (area under the curve; AUC), Total body clearance (CL), Volume of distribution (Vd)
TRPH-222 anti-drug antibodies (ADA) | Prior to treatment, prior to C3D1 and every 3rd cycle thereafter, EOT60
  Assess the incidence of subjects who develop ADA to the ADC with TRPH-222 monotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Hernandez- Ilizaliturri, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (7):
- United States (5):
  - Banner MD Anderson, Gilbert, Arizona
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No